CLINICAL TRIAL: NCT01358565
Title: Pharmacokinetics Of Orally Administered Fx-1006A In Subjects With Hepatic Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FX1A-105; B3461016
Record Dates: First submitted 2011-05-20; First posted 2011-05-23 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Mild Hepatic Dysfunction; Moderate Hepatic Dysfunction
MeSH Terms: interventions — tafamidis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mild and Moderate Hepatic Dysfunction (Active Comparator): Patients with mild and moderate hepatic dysfunction
  Interventions: Drug: Fx-1006A
- Healthy Volunteers (Active Comparator): Healthy volunteers
  Interventions: Drug: Fx-1006A

INTERVENTIONS:
Drug: Fx-1006A — A single oral 20 mg dose of Fx-1006A will be administered on Day 1 followed by 16 days of follow-up.
  Arms: Mild and Moderate Hepatic Dysfunction
Drug: Fx-1006A — A single oral 20 mg dose of Fx-1006A will be administered on Day 1 followed by 16 days of follow-up.
  Arms: Healthy Volunteers

SUMMARY:
This is a Phase I, open-label, single-dose study designed to assess the effects of hepatic dysfunction on the PK of orally administered Fx-1006A 20 mg soft gelatin capsules.

An adaptive 2-stage study design will be implemented. Initially (Stage 1), a group of 9 subjects with moderate hepatic dysfunction (Child-Pugh score of 7-9, inclusive) followed by a group of 9 healthy volunteer subjects with normal hepatic function who are comparable in age, gender, and weight to the hepatically impaired subjects will be enrolled to receive a single oral 20 mg dose of Fx-1006A each.

Data obtained from the first 2 groups will be analyzed and reviewed by the Sponsor to determine whether Fx-1006A PK is altered by hepatic dysfunction. If it is determined that hepatic dysfunction affects Fx-1006A PK, then Stage 2 will be commenced. During Stage 2, a group of 9 subjects with mild impairment (Child-Pugh score of 5-6, inclusive) will be enrolled to receive a single oral 20 mg dose of Fx-1006A each. Additional subjects with normal hepatic function may be enrolled to ensure appropriate demographic matching to the mild hepatically impaired subjects, with respect to age, gender, and weight.

During Screening, subjects will provide written informed consent to participate in the study and be reviewed against the study entrance criteria (including assessment of hepatic function) to determine eligibility. All subjects will provide blood and urine samples for clinical laboratory testing, drug testing, and pregnancy testing to determine eligibility.

Subjects who meet the entrance criteria during Screening will check in to the clinical site 1 day prior to dosing (Day 0) in the evening, and will be reviewed against the entrance criteria to confirm eligibility. Subjects will remain inpatient overnight for pre-dose assessments. Subjects will be fasted for a minimum of 8 hours prior to dosing the following day (water is allowed).

The single Fx-1006A dose will be administered on Day 1 under supervision of the Investigator or appropriate clinical site staff. Subjects will remain fasted for 4 hours after dosing (water is allowed) and will remain inpatient overnight for safety monitoring and PK sample collection.

Subjects will be discharged on Day 2, after they have completed the study procedures and the Investigator has determined that the subject is clinically stable. Subjects will return to the clinical site for out-patient visits on Days 3, 4, 6, 9, 12, and 16 for safety evaluations and PK sample collection. Day 16 will be the end of study visit.

ELIGIBILITY:
Inclusion Criteria:

All Subjects

* Subject is male or female (female subjects must be of non-child-bearing potential or willing to use a medically acceptable form of birth control during the study).
* Subject is between 18 to 70 years of age, inclusive.
* Subject is a cigarette smoker, consuming less than 15 cigarettes per day.
* Subject has given written informed consent.

Hepatic Dysfunction Subjects:

* Subject has hepatic dysfunction:

  1. Study Stage 1: Subject has moderate hepatic dysfunction (Child-Pugh score of 7-9, inclusive)
  2. Study Stage 2 (if commenced): Subject has mild hepatic dysfunction (Child-Pugh score of 5-6, inclusive)
* Subject's hepatic disease is deemed stable by the Investigator.
* Subject's pre-study clinical laboratory findings are within normal range or if outside of the normal range, deemed associated with underlying hepatic dysfunction or not clinically significant in the opinion of the Investigator and the sponsor.

Normal Hepatic Function Subjects:

* Subject is considered to be in good health in the opinion of the Investigator, as determined by:

  1. A pre-study physical examination with no clinically significant abnormalities
  2. Vital signs within normal ranges
  3. An ECG with no clinically significant abnormalities
* Subject's pre-study clinical laboratory findings are within normal range or if outside of the normal range not deemed clinically significant in the opinion of the Investigator and the Sponsor.

Exclusion Criteria:

* Subject has had a clinically significant illness in the four (4) weeks before screening.
* Subject shows evidence of a clinically significant underlying medical condition, including renal, cardiovascular, or metabolic dysfunction that, in the opinion of the Investigator, would represent a risk of study participation.
* Subject has any other clinically significant laboratory abnormality, as determined by the Investigator, within 21 days before dosing on Day 1.
* Subject has a history of clinically important disease that, in the opinion of the investigator, may put the subject at risk because of participation in this study.
* Subject is enrolled or plans to enroll in another clinical trial during this study or has received an investigational drug/device within 60 days before Day 1.
* Subject is known to be hepatitis B surface antigen (HbsAg) positive, anti-hepatitis C antibody (anti-HCV) positive, or human immunodeficiency virus (HIV) positive, or has any positive result during Screening.
* Subject has a history of alcohol abuse, or illicit drug use, physical dependence to any opioid, or drug abuse or addiction.
* Subject has a history of significant mental illness.
* Subject has positive urine drug screen test results within 21 days before Day 1, excluding alcohol. Alcohol consumption is not permitted within 72 hours before Day 1.
* Subject has a history of complications associated with providing blood samples.
* Subject reports donating greater than 150 mL of blood or donating plasma via plasmapheresis within 28 days prior to enrollment. All subjects will be advised not to donate blood for four weeks after completing the study.

Hepatic Dysfunction Subjects:

* Subject has an encephalopathy grade > 1.
* Subject has any clinically significant laboratory abnormality not associated with underlying hepatic impairment, as determined by the Investigator, within 21 days before dosing on Day 1.
* Unless being used to treat the subject's underlying hepatic disease, the subject has taken an over the counter (OTC) medication (including non-steroidal anti-inflammatory drugs (NSAIDs) or herbal preparations) within 48 hours before Day 1.

Normal Hepatic Function Subjects:

* Use of prescription medications in the 14 days prior to Day 1.
* Subject has taken an OTC medication (including NSAIDs or herbal preparations) within 48 hours before Day 1.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters are AUC0-last and Cmax | Daily

SECONDARY OUTCOMES:
Parameters are AUC0-inf, Cl, Tmax, t1/2; AUC, Cmax, and Cl will also be expressed in terms of unbound concentrations using the free fraction determined from protein binding assessments | Daily

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Newton Park, Port Elizabeth, South Africa

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=FX1A-105&StudyName=Pharmacokinetics%20Of%20Orally%20Administered%20Fx-1006A%20In%20Subjects%20With%20Hepatic%20Dysfunction